CLINICAL TRIAL: NCT06363253
Title: Understanding the Role of the Human Metagenome in Obesity, Metabolic Diseases, Chronic Inflammation, Sarcopenia and Sarcopenic Obesity - a Pilot Study
Brief Title: Pilot Study of the Human Metagenome in Metabolic Diseases
Status: Recruiting | Type: Observational
Sponsor: Sengkang General Hospital (Other)
Collaborators: Singapore General Hospital (Other); Lee Kong Chian School of Medicine, Nanyang Technological University (Unknown); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Chue Koy Min, Clinical Assistant Professor, Sengkang General Hospital
Other Study IDs: CIRB Ref: 2023/2073
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Sarcopenia; Sarcopenic Obesity; Chronic Inflammation; Metabolic Syndrome
Keywords: Obesity; Sarcopenia; Metabolic syndrome; Metagenomics; Metabolomics
MeSH Terms: conditions — Obesity; Sarcopenia; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal specimens; Salivary specimens; Mucosal specimens (these are samples with DNA, for aid in metagenomic sequencing to identify various microbial elements)
  Serum specimens; Urinary specimens (these are samples without DNA, for metabolite testing)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese: Patients with BMI > 27.5 kg/m2
  Interventions: Other: No specific intervention
- Sarcopenic: Patients who are sarcopenic, defined by the Asian Working Group on Sarcopenia 2014 criteria, which is defined as
  1. having low handgrip strength (<26kg for males; <18kg for females) AND/OR
  2. Low gait speed (<0.8m/s) AND
  3. Low muscle mass (<7.0kg/m2 for males; <5.7kg/m2 for females)
  Interventions: Other: No specific intervention
- Controls: Healthy volunteers who are not obese (BMI <27.5kg/m2), OR who are screened and found to not be sarcopenic
  Interventions: Other: No specific intervention

INTERVENTIONS:
Other: No specific intervention — Patient will undergo their routine clinical treatment for their related clinical condition (eg. anti-obesity or bariatric intervention for obese group; muscle strengthening interventions or necessary treatment for their concomitant medical condition for the sarcopenia group).
  Follow-up testing will include repeat assessment of the subjects metagenome and metabolome over time, and after intervention
  Control subjects will have no interventions performed as well.

SUMMARY:
This is a cohort study to understand the role of the human metagenome, and associated metabolites, in health and in various diseased states, in particular obesity as well as sarcopenia.

Recruited participants will have their fecal, salivary, urine, serum, and in certain instances, mucosal samples taken, for metagenomic sequencing and metabolite testing.

We hope to uncover various differences and signatures in the metagenome and metabolome in various diseased states, with potential future therapeutic applications in personalised medicine.

DETAILED DESCRIPTION:
The human metagenome comprises all nucleotide sequences isolated from all organisms living on and within an individual and has been shown to have significant alterations in relation to certain diseased states related to chronic inflammation, such as obesity and sarcopenia.

The gut bacteriome, and more recently the virome, has been shown to be significantly correlated with the obese phenotype, while gut microbiome dysbiosis is known to occur in individuals with sarcopenia. Clinically, there is an unmet clinical need to better personalize the treatment of patients with metabolic disorders such as obesity and metabolic syndrome, and patients suffering from sarcopenia and frailty as a result of aging. However, the literature regarding the metagenomic signatures associated with these disorders, in particular the non-bacteriome species, bacterial metabolites, and their relationship with host metabolism, were scarce.

Thus we hypothesize, that the human metagenome and metabolome, may play a role in influencing chronic inflammatory disorders related to metabolic disorders, such as obesity and diseases related to aging like sarcopenia and aging.

This is a cohort study, involving metagenomic sequencing and metabolomic analysis, of patients metagenome and metabolome, in various diseased states. A cohort of healthy control patients without obesity or sarcopenia will also be recruited.

Samples collected will include fecal, salivary, serum, urine, mucosal samples for metagenomic sequencing and metabolomic testing.

ELIGIBILITY:
Inclusion Criteria (obese cohort):

* Obese (BMI>27.5kg/m2)

Inclusion Criteria (sarcopenic cohort):

* Sarcopenic patients, defined as 1) low handgrip strength (<26 for males; <18kg for females), AND/OR low gait speed (<0.8m/s) AND low muscle mass (<7.0kg/m2 for males; <5.7kg/m2 for females)

Inclusion Criteria (control cohort):

- Healthy subjects without sarcopenia, and not obese (BMI<27.5kg/m2)

Exclusion Criteria:

* No informed consent
* Presence of intestinal stoma, hence inability to collect fecal samples

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese and sarcopenic patients will be recruited from patients from Sengkang General Hospital, opportunistically found during their management to be sarcopenic. Obese patients will be recruited from patients who are seen in the Sengkang General Hospital Weight Management Clinic.
  Controls are recruited from patients who are on follow-up for other non-related conditions found opportunistically to fit the inclusion criteria, as well as healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Metagenomic alterations | Period of 1 year
  Metagenomic alterations in the DNA/ RNA sequences of the saliva, stool (+/- mucosal) metagenome over time
Metabolomic alterations | Period of 1 year
  Changes in serum and urinary charged metabolites and small molecules over time

CONTACTS AND LOCATIONS:
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at the moment. Deidentified data can potentially be shared following institutional review board and hospital permission.